CLINICAL TRIAL: NCT05140278
Title: Convenience and Cost-aspects of a New 1-step Reconstitution Injectable Artesunate Compared to Conventional 2-step Injectable Artesunate for the Treatment of Severe Falciparum Malaria: a Multi-centre Study
Brief Title: Study to Compare Feasibility of 1-step Injectable Artesunate vs. Conventional 2-step Injectable Artesunate
Acronym: 1STEP-AS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Shanghai Fosun Pharmaceutical Industrial Development Co. Ltd. (Industry); University of Kinshasa (Other); National Institute for Medical Research, Tanzania (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MAL21006
Record Dates: First submitted 2021-11-17; First posted 2021-12-01 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2023-10

CONDITIONS: Severe Malaria
Keywords: Parenteral artesunate
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1-step Artesunate parenteral arm (Experimental): Argesun (Artesunate 60 mg)
  Interventions: Drug: Argesun 60mg (1 step parenteral artesunate)
- 2-step Artesunate parenteral arm (Experimental): Artesun (Artesunate 60 mg)
  Interventions: Drug: Artesun 60mg (2-step parenteral artesunate)

INTERVENTIONS:
Drug: Argesun 60mg (1 step parenteral artesunate) — Each vial of powder contains 60mg artesunate. Each ampoule of 6 ml solvent contains: sodium bicarbonate 8.4mg/ml; arginine 20mg/ml.
  Arms: 1-step Artesunate parenteral arm
Drug: Artesun 60mg (2-step parenteral artesunate) — Each vial of powder contains 60 mg artesunate. Each ampoule of 1 ml solvent contains 50 mg sodium bicarbonate. Each ampoule of 5 ml diluent contains 45 mg sodium chloride.
  Arms: 2-step Artesunate parenteral arm

SUMMARY:
The objectives of this study contains 3 parts: (1) a comparison of 1-step parenteral artesunate (AS) versus conventional 2-step parenteral artesunate in patients with severe malaria to assess the feasibility of administration, parasite and fever clearance times in two countries, (2) a quantification of convenience and costs of the new 1-step artesunate parenteral formulation versus the conventional formulation in a randomised study, (3) A cost analysis of 1-step parenteral artesunate using data from Part 1 & Part 2. This will assess health facility-level costs, and also health system costs to encompass all costs of a potential change from conventional to 1-step artesunate, including re-training, materials, and drug replacement.

The conventional formulation of injectable artesunate requires a 2-step reconstitution and dilution of the artesunate hemisuccinate powder. A new formulation of injectable artesunate has been developed by Fosun Pharma requiring a simpler 1-step reconstitution. Bioequivalence of the new formulation to the conventional formulation.

For part 1, a total number of participants of this study would be 200 participants, estimated 100 per site will be recruited. For part 2, a total number of 40 semi-structured interviews with study staff, health staff, policy makers, and stake holders; and survey/questionnaires with 150 health staff.

DETAILED DESCRIPTION:
Study design:

Part 1

A comparison of 1-step parenteral artesunate vs. conventional 2-step parenteral artesunate in patients with severe malaria to assess the feasibility of administration, parasite and fever clearance times of 1-step parenteral artesunate to conventional artesunate in 2 countries. Patients with severe malaria will be enrolled and randomly allocated to treatment with conventional injectable artesunate or 1-step injectable artesunate. A physical examination will be performed daily and every six hours on indication. Vital signs rec-orded hourly for unstable patients, then 6 hourly for stabilised patients, and at each follow-up visit. A symptom questionnaire will be taken daily to help identify adverse events. Patients will be asked to come back for a follow-up visit at day 7, 14, 21 and 28. Patients will not be followed up longer. In case of unresolved important sequelae at day 28, the patient will be followed and treated longer in order to provide the appropriate clinical care.

A Time and Motion study will record the time to prepare the artesunate solution for injection and administer treatment, number of actions performed to prepare treatment, and consumables used. Clinical, parasitological, and laboratory assessments will be recorded while patients are admitted in hospital and then weekly up to day 28 to assess recovery and determine final status.

Part 2

A mixed method social science study that entails semi-structure interviews and survey with study staff (involved in part 1), health workers (who treat severe malaria) and policymakers and stakeholders (who are involved in devising national malaria policy and its implementation), to assess the acceptability, feasibility, pros and cons, costs, and logistics and training implications of 1-step artesunate vs conventional artesunate. For both sites, semi-structure interviews will be conducted with minimum of a total of 40 respondents consisting of study staff, health staff and policy makers and stakeholders. The ultimate sample for semi-structure interviews will be dependent on the data saturation. For survey/questionnaire, a maximum number of relevant participants (study staff and health care staff) will be attempted to be recruited from two sites. A minimum of 150 study staff and health care staff will be recruited in the survey.

Part 3

A cost analysis of 1-step parenteral artesunate using data from Part 1 & Part 2. This will assess health facility-level costs, and also health system costs to encompass all costs of a potential change from conventional to 1-step artesunate, including re-training, materials, drug replacement.

In addition to time measurement, the observer will also record the resources used for the administration of artesunate. This will include the vials themselves, as well as other consumables required for the administration (syringes, needles, catheters, etc.).

Funder:

* Shanghai Fosun Pharmaceutical Industrial Development Co., Ltd
* Mahidol-Oxford Tropical Medicine Research Unit supported by the Wellcome Trust, UK (220211)

ELIGIBILITY:
Inclusion criteria

Part 1:

* Male and female children aged >3months and <16 years.
* Clinical diagnosis of severe P. falciparum malaria; or parasitological confirmed P. falciparum hyperparasitaemia >350,000/ uL.
* Positive malaria test result, by rapid diagnostic test RDT.
* Weight of 5 kg or greater.
* Written informed consent by the parent or guardian.

Part 2:

Study staff and health staff

* Study staff who prepare and administer Artesunate injection to patients in the study or health staff who have not administer the Artesunate injection to patients in the study by themselves but are either aware of malaria treatment, Artesunate injection, or have observed the treat-ment provided to severe malaria patients.
* Written informed consent by the study staff and health staff

Study staff for a short video-record

* Study staff who would like to participate in the video record of a procedure to show how 1-step and 2-step Artesunate injections are prepared and administered.
* Written informed consent by the study staff

Policymakers and stakeholders

* Those who are working in the National Malaria Control Program (NMCP) or relevant organizations (WHO, INGOs/NGOs) within the country.
* Written informed consent by the potential participant

Exclusion criteria

Part 1:

* Participation in other intervention studies
* Known allergy to artemisinin derivatives.
* Known history of parenteral treatment for severe malaria for the current episode of illness before admission. Treatment before admission with an oral antimalarial drug (used for the treatment of uncomplicated malaria) or a single dose of pre-referral rectal artesunate are not exclusion criteria.

Part 2:

Study staff and health staff; Policymakers and stakeholders; Study staff and health staff for a short video-record

* Unwilling to participate in the study
* Unable to communicate

Ages: 3 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2022-07-18 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2023-08-11 (Actual)

PRIMARY OUTCOMES:
Time to administration of treatment comparing 1-step vs. conventional 2-step parenteral artesunate formulations | 3 days
  Time to administration of treatment comparing 1-step vs. conventional 2-step parenteral artesunate formulations (by time-and-motion methods).
Costs of administration of 1-step vs. conventional 2-step parenteral artesunate formulations | 3 days
  Costs of administration of 1-step vs. conventional 2-step parenteral artesunate formulations at health facility, and at health system level.

SECONDARY OUTCOMES:
Implementation perspective assessment of 1-step formulation of parenteral artesunate | 45 minutes
  Implementation perspective assessment of 1-step formulation of parenteral artesunate by interview study staff, health staff, and policymakers and stakeholders
Practicability assessment of 1-step formulation of parenteral artesunate | 45 minutes
  Practicability assessment of 1-step formulation of parenteral artesunate by interview study staff, health staff, and policymakers and stakeholders
Satisfaction assessment of 1-step formulation of parenteral artesunate | 45 minutes
  Satisfaction assessment of 1-step formulation of parenteral artesunate by interview study staff, health staff, and policymakers and stakeholders

OTHER OUTCOMES:
Parasite clearance half-life and other parasite clearance parameters compared between 1-step vs. conventional 2-step parenteral artesunate formulations. | 28 days
  Parasite clearance half-life and other parasite clearance parameters (PC50, PC90, 12-hour parasite reduction ratio) compared between 1-step vs. conventional 2-step parenteral artesunate formulations.
Time from start parenteral treatment to follow up treatment with an oral ACT | 28 days
  Time from start parenteral treatment to follow up treatment with an oral ACT (recovery to per os treatment) of 1-step vs. conventional 2-step parenteral artesunate formulations.
Fever clearance time | 28 days
  Fever clearance time (i.e. the time taken for the tympanic temperature to fall below 37.5˚C and remain there for at least 24 hours) of 1-step vs. conventional 2-step parenteral artesunate formulations
Incidence of adverse events | 28 days
  Incidence of adverse events by study arms within the first 28 days.
Incidence of serious adverse events by study arms | 28 days
  Incidence of serious adverse events by study arms

CONTACTS AND LOCATIONS:
Overall Officials: Caterina Fanello, Ph D, Principal Investigator — Kinshasa School of Public Health; Samwell Gesase, MD, Principal Investigator — Magunga District Hospital; Arjen Dondrop, MD, Principal Investigator — Mahidol Oxford Tropical Medicine Research Unit Bangkok, Thailand; Marie Akatshi Onyamboko, Principal Investigator — Kinshasa School of Public Health, University of Kinshasa, DRC
Locations (1):
- KIMORU (KIMORU /ESP Research Center), Kinshasa, Democratic Republic of the Congo

IPD SHARING:
Plan to Share IPD: Yes
Participant's data and results from blood analyses stored in the database may be shared according to the terms defined in the MORU data sharing policy with data repositories or other researchers to use in the future. All personal information will be de-identified so that no individual can be identified from their treatment records, through interviews.
URL: https://www.tropmedres.ac/units/moru-bangkok/bioethics-engagement/data-sharing

DOCUMENTS (2):
  • Study Protocol (2021-08-18): https://cdn.clinicaltrials.gov/large-docs/78/NCT05140278/Prot_002.pdf
  • Statistical Analysis Plan (2023-08-23): https://cdn.clinicaltrials.gov/large-docs/78/NCT05140278/SAP_003.pdf